CLINICAL TRIAL: NCT05599087
Title: Encapsulated Acellular System From Mesenchymal Stem Cells for Endodontic Treatment of Patients With Apical Periodontitis: Phase I Clinical Trial.
Brief Title: Encapsulated Acellular System From Mesenchymal Stem Cells for Dental Pulp Regeneration
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: Cells for Cells (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAndes2
Record Dates: First submitted 2022-10-25; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Periapical Periodontitis
Keywords: mesenchymal stem cells; regenerative procedures; dental pulp; pulp regeneration; allogenic acellular system
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acellular system (Experimental): Regenerative Endodontic Procedure (REP) the acellular system derived from umbilical cord-derived mesenchymal stem cells encapsulated in a platelet-poor plasma-derived biomaterial.
  Interventions: Biological: Acellular system

INTERVENTIONS:
Biological: Acellular system — Regenerative Endodontic Procedure Tissue engineering procedure

SUMMARY:
To evaluate the security and efficacy in the administration of encapsulated acellular system derived from Mesenchymal Stem Cells as a novel regenerative endodontic procedure which to promote the pulpar regenration.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients (ASA I).
* Patient presenting with a maxillary or mandibular incisor/canine and mandibular premolar with mature apex, pulpal necrosis, and apical radiographic evidence of apical periodontitis (PAI ≥2 and CBCTPAI ≥1).
* Patient presents with a tooth that does not respond to electrical and thermal pulp testing.
* Patients with restorable teeth (considering the definition of class A or B, according to Samet and Jotkowitz classification) without the need for a single fine prosthesis (crown) or major restoration.

Exclusion Criteria:

* Patients not available for the follow-up period (27 weeks).
* Patients who will undergo orthodontic treatment in the next six months.
* Patients with reports of allergies to any material or medication used in the study.
* Pregnant patients.
* Heavy smokers (more than 10 cigarettes per day).
* Patients with a history of systemic diseases that impair immune function, such as diabetes mellitus, immunodeficiency, leukemia, Addison's and Cushing's disease.
* Patients who have used immunosuppressive drugs or chemotherapy, 3 months before the study. Or that they will be irradiated or undergo chemotherapy.
* Patients who have endodontically treated teeth.
* Patients who have teeth with signs of severe root resorption.
* Patients who have teeth with mobility class III or Dens invaginatus.
* Patients who have teeth with a history of avulsion-type dentoalveolar trauma.
* Patients who have teeth with clinical and/or radiographic evidence of root fracture.
* Patients who have teeth that cannot be completely isolated with rubber dam.
* Patients who have teeth with more than one root or root canal.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-12-30 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Regeneration of dental pulp | 6 months
  Patients are expected to have a decrease in the size of the periapical lesion in some of the three dimensions, or an increase of no more than 0.1 mm in one of them, when evaluating radiographic and cone beam computed tomography (CBCT) .

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de los Andes, Las Condes, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided